CLINICAL TRIAL: NCT01566084
Title: Efficacy of Dietary Sodium Restriction of Improving Vascular Endothelial Function in Middle Aged and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Douglas Seals, College Professor of Distinction, University of Colorado, Boulder
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: B5114; F31AG033994 (NIH)
Record Dates: First submitted 2012-03-23; First posted 2012-03-29 (Estimated); Results first posted 2014-06-20 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal sodium (Other): Subjects on a 1200 mg sodium diet are given 2300 mg sodium in the form of slow sodium tablets to bring them back up to a normal salt intake. Subjects then cross-over to the low sodium condition in the second half of the study.
  Interventions: Drug: Slow sodium tablets
- Low sodium (Other): Subjects on a 1200 mg salt diet are given placebo pills in order to maintain them on a low salt diet. Subjects then cross-over to the normal sodium condition in the second half of the study.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Slow sodium tablets — The normal salt condition is maintained with 2300 mg / day in the form of slowly released salt (NaCl) tablets.
  Arms: Normal sodium
Other: placebo — Placebo tablets are administered to maintain the low sodium condition.
  Arms: Low sodium

SUMMARY:
The investigators hypothesize that reducing salt in the diet will improve the function of blood vessels in middle aged and older adults with moderately elevated systolic blood pressure, by increasing the amount of BH4 and nitric oxide in your blood vessels and reducing the amount of oxidative stress.

DETAILED DESCRIPTION:
The improvement in blood vessel function will be determined over a 10 week period. Subjects will be randomly assigned to either a 'low salt' condition (placebo pills + 1200 mg dietary sodium) or a 'normal salt' condition (2300 mg sodium chloride pills + 1200 mg dietary sodium) and monitored for 5 weeks. After the initial set of 5 weeks, the subjects are switched into the opposite condition, completing the cross-over study design. During weeks 1-4 and 6-9, subjects are monitored weekly with 24 hour urine collections and diet logs. The assessment of the primary outcome (blood vessel function) is completed during weeks 5 and 10. BH4 and ascorbic acid are also administered during weeks 5 and 10 to measure the effects of sodium intake on endogenous BH4 levels and vascular oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* 50-79 years of age
* SBP 130-159 mmHg

Exclusion Criteria:

* Have been sick with an infection in the past two weeks
* Are currently sick or have ongoing health problems such as kidney or CVD
* Have lost more than 11 lbs. in the last 3 months
* Are taking any type of antioxidants
* Smoke or have alcohol problems
* Have blood glucose levels higher than 126 mg/dL
* Have resting SBP below or less than 100 mmHg or greater than 159 mmHg
* Have a resting diastolic blood pressure greater than 99 mmHg
* Have a BMI greater than 40 kg/m^2
* Are presently consuming less than 9 or greater than 18 grams of salt / day
* Have a baseline FMD of greater than 6%
* Are taking any of the following types of drugs: blood thinners, anti-seizure medications, ant-inflammatory drugs
* Participate in any high endurance athletic training
* Taking Hormone Replacement Therapy
* Have not been post-menopausal for at least 1 year

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen L Jablonski, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- Clinical Translational Research Center, Boulder, Colorado, United States

REFERENCES:
- See also: Integrative Physiology of Aging Laboratory Website — http://www.colorado.edu/intphys/research/cardiovascular.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Slow Sodium Tablets (Start): Subjects on a 1200 mg sodium diet are given 2300 mg sodium in the form of slow sodium tablets to bring them back up to a normal salt intake.
  Subjects then cross over to the opposite condition in the second half of the study.
- Placebo: Subjects on a 1200 mg salt diet are given placebo pills in order to maintain them on a low salt diet.
  Subjects then cross over to the opposite condition in the second half of the study.
Period: Overall Study
Arm/Group | Slow Sodium Tablets (Start) | Placebo
Started | 7 | 10
Completed | 7 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 11 Men and 6 post-menopausal women were enrolled.
Groups:
- Slow Sodium Tablets (Start): Subjects on a 1200 mg sodium diet are given 2300 mg sodium in the form of a slow sodium tablets to bring them back up to a normal salt intake. This is administered through 10 tablets day.
  Subjects then cross-over to the placebo arm in the second half of the study.
- Placebo (Start): Subjects on a 1200 mg salt diet are given placebo pills in order to maintain them on a low salt diet.
  Subjects then cross over to the slow sodium tablet arm in the second half of the study.
- Total: Total of all reporting groups
Arm/Group | Slow Sodium Tablets (Start) | Placebo (Start) | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (7) | 62 (7) | 62 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Improved Flow Mediated Dilation
Description: FMD is analyzed at weeks 5 and 10 or after each condition in this cross-over study design. Subjects are randomly assigned to a low salt or normal salt condition for the first set of 5 weeks and then crossed over to the other condition for the second set of 5 weeks.
Time Frame: Week 5 (after first condition of low salt or normal salt), Week 10 (after second condition, opposite to first)
Population: All subjects are analyzed under each condition because of the cross-over design.
Measure: Mean (Standard Deviation); unit: percentage dilation
Groups:
- Normal Sodium Diet: Subjects on a 1200 mg sodium diet are given 2300 mg sodium in the form of a salt pill to bring them back up to a normal salt intake.
- Low Sodium Diet.: Subjects on a 1200 mg salt diet are given placebo pills in order to maintain them on a low salt diet.
Arm/Group | Normal Sodium Diet | Low Sodium Diet.
Number analyzed (Participants) | 17 | 17
percentage dilation | 3.57 (1.59) | 6.01 (2.31)

2. Secondary Outcome: Vascular Oxidative Stress
Description: Change in FMD following acute infusion of ascorbic acid (a dose known to scavenge superoxide) is measured at the end of 5 weeks of sodium condition (low and normal intake) as an index of vascular oxidative.
Time Frame: Immediately following acute infusion of ascorbic acid on Weeks 5 and 10
Population: Ascorbic acid is missing in one participant due to a failed i.v.
Measure: Mean (Standard Deviation); unit: percentage dilation
Groups:
- Normal Sodium Saline; Normal Sodium Ascorbic Acid; Low Sodium Ascorbic Acid: Subjects on a 1200 mg sodium diet are given 2300 mg sodium in the form of slow sodium tablets to bring them back up to a normal salt intake.
  FMD is assessed following an acute supraphysiological infusion of ascorbic acid (known to scavenge superoxide) compared to an equal volume of normal saline.
- Low Sodium Saline: Subjects on a 1200 mg salt diet are given placebo pills in order to maintain them on a low salt diet.
  FMD is assessed following an acute supraphysiological infusion of ascorbic acid (known to scavenge superoxide) compared to an equal volume of normal saline.
Arm/Group | Normal Sodium Saline | Low Sodium Saline | Normal Sodium Ascorbic Acid | Low Sodium Ascorbic Acid
Number analyzed (Participants) | 17 | 17 | 16 | 16
percentage dilation | 3.57 (1.69) | 6.01 (2.31) | 4.90 (2.84) | 5.51 (2.36)

3. Secondary Outcome: BH4 Bioavailability
Description: Change in FMD following acute oral tetrahydrobiopterin (BH4) is measured at the end of 5 weeks of sodium condition (low and normal intake) as an index of BH4 bioavailability.
Time Frame: Immediately following acute administration of BH4 on Weeks 5 and 10
Population: BH4 could not be administered to 3 participants due to canceled visits.
Measure: Mean (Standard Deviation); unit: percentage dilation
Groups:
- Normal Sodium Placebo; Normal Sodium BH4; Low Sodium BH4: Subjects on a 1200 mg sodium diet are given 2300 mg sodium in the form of slow sodium tablets to bring them back up to a normal salt intake.
  FMD is assessed following acute oral tetrahydrobiopterin (BH4) or placebo is measured at the end of 5 weeks of sodium condition (low and normal intake) as an index of BH4 bioavailability.
- Low Sodium Placebo: Subjects on a 1200 mg salt diet are given placebo pills in order to maintain them on a low salt diet.
  FMD is assessed following acute oral tetrahydrobiopterin (BH4) or placebo is measured at the end of 5 weeks of sodium condition (low and normal intake) as an index of BH4 bioavailability.
Arm/Group | Normal Sodium Placebo | Low Sodium Placebo | Normal Sodium BH4 | Low Sodium BH4
Number analyzed (Participants) | 17 | 17 | 14 | 14
percentage dilation | 3.57 (1.69) | 6.01 (2.31) | 5.78 (2.02) | 6.11 (2.32)

ADVERSE EVENTS:
Groups:
- Normal Sodium: Subjects on a 1200 mg sodium diet are given 2300 mg sodium in the form of slow sodium tablets to bring them back up to a normal salt intake.
- Low Sodium: Subjects on a 1200 mg salt diet are given placebo pills in order to maintain them on a low salt diet.
Arm/Group | Normal Sodium | Low Sodium
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
Due to the complexity, burden, and, in some cases, invasiveness of the study design and procedures, only a limited number of subjects could be studied.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No